CLINICAL TRIAL: NCT03424902
Title: Study of New Predictors and Short Term Outcomes of Paravalvular Leakage Post Transcatheter Aortic Valve Implanation
Brief Title: Study of New Predictors and Short Term Outcomes of Paravalvular Leakage After Transcatheter Aortic Valve Implanation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marwan Sayed Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Marwan Sayed Mahmoud, Assiut university hospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 13254
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Paravalvular Leakage After TAVI
MeSH Terms: interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: patients with no or mild paravalular leakage
  Interventions: Diagnostic Test: cardiac computed tomography and cardiac catheterization
- group 2: patients with moderate or or severe paravalvular leakage
  Interventions: Diagnostic Test: cardiac computed tomography and cardiac catheterization

INTERVENTIONS:
Diagnostic Test: cardiac computed tomography and cardiac catheterization — assesment of certain predictors with CT and fluroscopy for paravalvular leakage

SUMMARY:
The presence of aortic regurgitation (AR) jet from the aorta into the left ventricle is the most common complication after TAVI, occurring in about 70% of patients but usually trivial or mild (4, 5). In most previous studies, mild AR was not associated with a significantly shorter survival time (4, 5); however, the PARTNER trial demonstrated that it may be associated with worse long-term prognosis (3).

Significant AR (moderate and severe) is less common, occurring in approximately 15-20% of cases(6), and is considered one of the most important prognostic factors of mortality during short- and long-term follow-up (7, 8). It is, therefore, essential to understand the mechanisms and risk factors associated with the occurrence of AR in order to minimize its incidence .

Significant PVL most commonly results from(9):

1. Incomplete prosthesis apposition to the native annulus due to calcification or annular eccentricity
2. undersizing of the device and/or
3. malpositioning of the valve . These observations seem to be true for both balloon-expandable and self-expandable THVs.

However there are some new predictors which may correlate to occurance of paravalvular leakage including :

1. Eccentricity of aortic valve calcification.
2. Characterization of aortic annular calcification.
3. Associated mitral annular calcification.
4. Angle of LVOT to ascending aorta measurement (LVOT-AO).
5. The depth of implantation of valve in relation to aortic cusps.

DETAILED DESCRIPTION:
Aim of work Assessment of new predictors and short term outcomes of paravalvular leakage after transcatheter aortic valve implantation (TAVI).

These new predictors are :

* Eccentricity of aortic valve calcification.
* Characterization of aortic annular calcification.
* Mitral annular calcification.
* Angle of LVOT to ascending aorta measurement (LVOT-AO).
* The depth of implantation of valve in relation to aortic cusps Patients and methods. The study will include ( ) patients both retrospective and prospective observational study

Inclusion criteria :

The following will be eligible for TAVI :

1. Intermediate or high risk patient for surgical aortic valve replacement (SAVR) STS/EuroSCORE II >4% or logistic EuroSCORE I >10%(10).
2. Contraindications for open chest surgery, such as(10) :

   1. Expected high perioperative risk due to comorbidities not adequately reflected by scores :

<!-- -->

1. Procelain aorta
2. Squelae of chest radiation.
3. Severe chest deformation or scoliosis.
4. Previous cardiac surgery .

Exclusion criteria(10) :

A-clinical conditions.

1. active endocarditis,
2. myocardial infarction within 14 days
3. cardiogenic shock
4. Life expectancy of less than 1 year

B-Anatomical conditions:

1. short distance between coronary ostia and aortic valve annulus.
2. Size of aortic annulus out of range for TAVI(range from 18mm - 27mm)(10).

C-Associated cardiac condition requiring concomitant intervention eg severe CAD require CABG ,aneurysm of ascending aorta ,severe mitral or tricuspid valve disease.

All patient will undergo :

1. Written consent.
2. Detailed history including symptoms (NYHA class) ,co morbidities(diabetes ,hypertension ,ischemic heart disease,previous PCI ,renal impairment,peripheral arterial disease , chronic obstructive pulmonary disease,cerebrovascular disease ,atrial fibrillation ,..)
3. Clinical examination
4. Electrocardiogram(detection of conduction disturbance , ischemic changes).
5. Laboratory investigation (hemoglobin level ,creatinine,glomerular filteration rate(GFR))
6. Echocardiography(11) :

1-Assesment of aortic valve by

1. Mean and maximum pressure gradiant .
2. Aortic valve area by continuity equation.
3. Measurement of aortic valve annulus(by both transthoracic echocardiography in parasternal long axis view and transesophgeal echocardiography in long axis view ) .
4. Assesment of associated aortic regurge (regurge jet,regurge fraction and volume) 2- Assesment of EF(by M-mode and simpsons method). 3-Assesment of other valves . 7-Computed tomography (cardiac CT )

<!-- -->

1. Annular dimensions. Two diameters, the anteroposterior (AP) short axis and the mediolateral (ML) long axis will be measured, and the mean ([ML plus AP] divided by 2) will be calculated(12).

   The Cover Index is defined as 100x(nominal prosthesis diameter - CT mean annulus Diameter)/nominal prosthesis diameter (13,14), and the

   Eccentricity Index was calculated as 100 x(1 -(aortic annulus minimum diameter /maximum diameter) (15).
2. Annular calcium . The cross-sectional axial annulus plane is used for the following analysis:

   1-Amount of calcium is measured using Agatston calcium score(AgS)(16). 2-Characterization of annular calcification : Annular calcification is measured in two planes, depth (D) and width (W), and evaluated for shape (1 for protruding [D>W], 2 for round [D=W], and 3 for adherent [W>D]) for each side (noncoronary, right coronary, and left coronary annulus side)(12).
3. Eccentricity of aortic valve calcification(EoC):

   The EoC is defined as the maximum absolute difference in calcium volume scores between 2 adjacent sectors (bi-partition method) or between sectors based on leaflets (leaflet-based method) (16).
4. Angle of LVOT to ascending aorta measurement (LVOT-AO). We consider the angle between the axis of the first 4 cm of the ascending aorta representing the contact surface with the upper part of the bioprosthesis and the LVOT axis representing the landing zone of the prosthesis. . This angle is determined on CT or using left ventriculography in RAO 30° during preparation of the patients for the procedure (17).
5. Mitral annular calcification:

   is qualitatively determined by circumferential involvement of mitral ring, mild =less than 1/3 of mitral annulus , moderate =between 1/3and 1/2 of mitral annulus , severe =calcification more than half mitral annulus circumference (20).

   TAVI procedure:

   The detailed steps of procedure are reported by Nijhoff F,etal (19) .TAVI is performed through transfemoral or transapical approach, based on the feasibility of the iliofemoral anatomy and suitable access sites. All procedures are performed in a fully equipped hybrid cardiac catheterization laboratory. Surgical cutdown or suture-mediated closure device are used to close the vascular access site at the femoral arteries.

   Transesophageal echocardiography is used to support TAVI procedures, and fluoroscopy is used to guide the deployment of the valves and prosthesis positioning. Both predilatation of the native valve and prosthetic valve implantation are performed during rapid right ventricular pacing (160 to 200 beats/min) (19). Prosthesis position, function, and coronary ostia patency are assessed with transesophageal echocardiography and fluoroscopy .

   Procedural factors which relate to paravalvular leakage include:
   1. Valve type (balloon expandable or self expandable).
   2. Valve size in relation to aortic annulus size (cover index).
   3. The depth of implantation of valve in relation to aortic cusps.

   Depth of final device position in the LVOT will be measured using a final aortogram of the deployed bioprosthesis in RAO projection, displaying the aortic valve in optimal alignment with all 3 leaflets visible in the same plane. The depth of delivery is defined as the distance from the native aortic annular margin on the side of the non coronary cusp (NCC) to the most proximal edge on the corresponding side (deepest in the left ventricle) of the deployed stent-frame .In addition, the depth of delivery from the annular margin of the left coronary cusp to the corresponding side will be measured(20).

   Assesment of paravalvular leakage :

   1-Angiographic evaluation of paravalvular leakage Ten minutes after the deployment of the prosthetic valve, angiography of the aortic root is performed to assess the severity of aortic regurgitation according to Sellers criteria (21).

   (0) no regurgitation.

   (1) only trace of contrast could be seen in the left ventricle, and it is cleared in each systole.

   (2) contrast filling the entire LV in diastole with less density compared with opacification of the ascending aorta.

   (3) contrast filling the entire LV in diastole equal in density to the contrast opacification of the ascending aorta.

   (4) contrast filling of the entire LV in diastole on the first beat with greater density compared with the contrast opacification of the ascending aorta.

   Two observers independently score the images. In case of discrepancy the images will be re-evaluated and consensus will be reached by a third observer.

   2-Intraprocedural Transesophageal echocardiography : Both 2D and 3D TEE will be used to assess origin and severity of paravalvular leakage during procedure.

   3-Transthoracic Echocardiographic study:

   All patients will be evaluated after TAVI by pre-discharge transthoracic echocardiography. The extent of PVL is assessed according to the main VARC criteria(9):

<!-- -->

1. Semiquantitative parameters

   1-Diastolic flow reversal in the descending aorta-pulsed wave : mild (Absent or brief) ,moderate ( early diastolic Intermediate), severe (Prominent holodiastolic) 2-Circumferential extent of prosthetic valve paravalvular regurgitation: (0) no regurgitation; (1) mild PVL is defined as<10 % circumferential extent; (2) moderate PVL was defined as [>10 % but<30 % of PVL and (3) severe PVL is defined as >30 % according to the updated VARC guideline , that is the circumferential extent of PVL in a parasternal short-axis view (19).
2. Quantitative parameters:

   1. Regurgitant volume (ml/beat) mild (<30) , moderate (30-59) ,severe (>60).
   2. Regurgitant fraction (%) mild (< 30), moderate (30-49) ,severe (>50).
   3. Effective regurgitant orifice area (cm2) mild (<0.10) ,moderate (0.10-0.29) , severe (>0.30).

      Follow up patients after 1month :

   <!-- -->

   1. Clinical follow up (symptoms,hospital readmission ).
   2. Echocardiographic reassessment of paravalvular leakage using the VARC criteria .

Statistical analysis The collected data will be tabulated and statistically analyzed and will be shown in tables and figures.

ELIGIBILITY:
Inclusion Criteria:

* The following will be eligible for TAVI :

  1. Intermediate or high risk patient for surgical aortic valve replacement (SAVR) STS/EuroSCORE II >4% or logistic EuroSCORE I >10%(10).
  2. Contraindications for open chest surgery, such as(10) :

     1. Expected high perioperative risk due to comorbidities not adequately reflected by scores :

  <!-- -->

  1. Procelain aorta
  2. Squelae of chest radiation.
  3. Severe chest deformation or scoliosis.
  4. Previous cardiac surgery .

Exclusion Criteria:

* A-clinical conditions.

  1. active endocarditis,
  2. myocardial infarction within 14 days
  3. cardiogenic shock
  4. Life expectancy of less than 1 year

B-Anatomical conditions:

1. short distance between coronary ostia and aortic valve annulus.
2. Size of aortic annulus out of range for TAVI(range from 18mm - 27mm)(10).

C-Associated cardiac condition requiring concomitant intervention eg severe CAD require CABG ,aneurysm of ascending aorta ,severe mitral or tricuspid valve disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -Intermediate or high risk patient for surgical aortic valve replacement (SAVR) STS/EuroSCORE II >4% or logistic EuroSCORE I >10%
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of significant paravalvular leakage | 1 .5 year
  moderate or severe